CLINICAL TRIAL: NCT05841914
Title: DECODE VRL - Multicentric Implementation and Clinical Validation of Standardized, Innovative Molecular Diagnostics for VitreoRetinal Lymphoma
Brief Title: Multicentre Implementation and Validation of a Molecular Diagnostic for VitreoRetinal Lymphoma
Acronym: DecodeVRL
Status: Recruiting | Type: Observational
Sponsor: Vinodh Kakkassery, MD (Other)
Collaborators: University Hospital Tuebingen (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor-Investigator, Vinodh Kakkassery, MD, PD Dr. med, principal investigator, University of Luebeck
Organization: University of Luebeck (Other)
Other Study IDs: 70114881
Record Dates: First submitted 2023-04-02; First posted 2023-05-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Vitreoretinal Lymphoma
Keywords: Vitreoretinal lymphoma; primary CNS lymphoma; improved detection; molecular diagnostics; diagnostic standardisation; health services research; prospective study
MeSH Terms: conditions — Intraocular Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vitreous aspirates, Anterior chamber water samples, whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to gain new insights into the changes in proteins, genes and other molecular biological substances in the aqueous humour, vitreous humour, blood serum and, in rare cases, retina/choroid samples in patients with ocular lymphoma disease. The hope is that this will expand the understanding of the mechanisms of the disease and thus contribute to improved and simplified diagnosis and treatment strategies in the future. The aim is the inclusion of at least 220 patients during the study period. The main questions it aims to answer are:

* to evaluate the diagnostic quality of extended molecular diagnostics (based on standard work-up) of vitreous samples for the specific VitreoRetinalLymphoma (a type of ocular lymphoma disease) diagnosis in comparison to standard work-up alone.
* To monitor VRL patients as part of regular tumour follow-up over a period of 24 months to determine the value of biomarkers with regard to treatment response and development of recurrence in the eye. Similarly, the vitritis patients are followed up by telephone every six months for a period of 24 months, during which questions of any interim occurrence of a VRL or other cancerous tumors are asked according to a defined catalogue of questions.

DETAILED DESCRIPTION:
Vitreoretinal lymphoma (VRL) is a rare intraocular neoplasm that is considered a variant of primary CNS lymphoma (PCNSL) and may manifest primarily or secondarily in the vitreous and retina. The distinction between vitritis/uveitis and VRL is clinically difficult and requires cytological examination of invasively obtained vitreous material for definitive diagnosis. Due to the time-consuming material collection and the clinical masquerade as vitritis, there are often significant delays in diagnosis. In addition, only a few centres have sufficient experience in the diagnosis and therapy of this rare lymphoma entity. The sensitivity of established tests (cytology, immunophenotyping, clonality analysis) on vitrectomy specimens is at most 70% for VRL. A standardised diagnostic procedure has not yet been defined.

This study aims to implement a network for standardised molecular analysis of VRL, to evaluate the impact of standardised molecular diagnostics on diagnostic quality prospectively through clinical follow-up.The network partners will prospectively send diagnostic vitreous samples from patients with suspected VRL, process them centrally in a standardised manner and subject them to multiparametric molecular diagnostics (mutation analysis and clonality detection using next generation sequencing, miRNA analysis). Due to the rarity of the disease, a recruitment period of 4 years is planned with the inclusion of at least 220 patients with suspected VRL, including 50 in whom VRL can ultimately be confirmed. At the time of surgery, the diagnostic chain (including type and duration of symptoms, clinical course up to vitrectomy) will be evaluated using questionnaires and a qualitative interview with stakeholders (patients, ophthalmologists, pathologists, oncologists). In order to validate the quality of molecular diagnostics and to evaluate the significance for the course of the disease (treatment failure, local recurrence, CNS involvement and recurrence), a prospective clinical documentation of the course of the disease with an observation period of 2 years for VRL patients is being carried out in cooperation with the CNS Lymphoma Working Group of the German Lymphoma Alliance.

Analogous to the VRL patients, the vitritis patients are asked by telephone every six months for two years whether they have been diagnosed with VRL or PCNSL. All VRL patients will be included in a clinical registry. Remaining biomaterial from vitreous bodies will be deposited in a central biobank for future research projects and biomarker establishment, independent of diagnosis.

The aim of the project is to implement a standardised and quality-assured molecular genetic analysis of VRL in specialised centres throughout Germany and thus to achieve an improved and more time-efficient diagnosis of this rare and aggressive disease. The network for the diagnosis of VRL and the clinical registry can also serve as a basis for the development of therapy studies in the future in cooperation with the CNS Lymphoma Working Group of the German Lymphoma Alliance, which is largely lacking in this entity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of the presence of VRL with indication for diagnostic vitrectomy. Clinical suspicion is based on the assessment of the treating physicians in the clinics participating in this study.
* Age over 18 years.
* Written informed consent to participate in the study.

Exclusion Criteria:

* Systemic chemotherapy for lymphoma within 3 months prior to vitrectomy.
* Cortisone use within 2 weeks before vitrectomy, macular oedema, posterior synechiae, rubeosis iridis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical suspicion of vitreoretinal lymphoma
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
To implement a standardised diagnostic work-up of vitreous samples from patients with suspected VRL | 6 years
  The diagnostic work-up would be from patients with suspected VRL including NGS-based mutation and B-cell clonality analysis and quantification of miRNAs 19b, 21 and 92 for the participating ophthalmology centres.
Rate of correct diagnosed VRL and vitritis with the use of extended molecular diagnostics versus standard work-up alone | 6 years
  The evaluation of the diagnostic sensitivity and specificity of extended molecular diagnostics (based on standard work-up) of vitreous samples for VRL diagnosis in comparison to standard work-up alone.
Rate of patients with VRL or vitritis within the follow up of 24 Months after diagnostics | 24 Months for each patient, all in all a 6 year frame for all patients.
  Follow-up of VRL patients during regular tumour follow-up over a period of 24 months to determine the predictive significance of the biomarkers with regard to therapy response, development of recurrence in the eye, second eye involvement as well as CNS involvement and recurrence. Similarly, the vitritis patients are followed up by telephone every six months for a period of 24 months, during which any interim occurrence of a VRL or a PCNSL as well as further questions are asked according to a defined catalogue of questions.

SECONDARY OUTCOMES:
Establish a central VRL clinical registry | 6 years
  A central VRL clinical registry should be established to facilitate the exchange of information. The registry will be established with the support of the German Lymphoma Alliance and Retina.net.
A Biobank of VRL and Vitritis from residual material | 6 years
  Establishment of a residual material biobank (especially DNA and RNA) of VRL and the control group vitritis.

CONTACTS AND LOCATIONS:
Overall Officials: Vinodh Kakkassery, PD Dr.med., Study Chair — University of Luebeck
Locations (1):
- University Clinic of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany